CLINICAL TRIAL: NCT01053494
Title: The TOUCH Project: Reducing Distress and Promoting Quality of Life Via Caregiver Massage of Children Undergoing Treatment for Cancer
Brief Title: Massage Therapy Given by Caregiver in Treating Quality of Life of Young Patients Undergoing Treatment for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00011619; NCI-2009-01456 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97709 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Undifferentiated Leukemia; Angioimmunoblastic T-cell Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Burkitt Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Mantle Cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Essential Thrombocythemia; Extramedullary Plasmacytoma; Intraocular Lymphoma; Isolated Plasmacytoma of Bone; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Meningeal Chronic Myelogenous Leukemia; Noncontiguous Stage II Mantle Cell Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Primary Myelofibrosis; Primary Systemic Amyloidosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Stage 0 Chronic Lymphocytic Leukemia; Stage I Childhood Anaplastic Large Cell Lymphoma; Stage I Childhood Hodgkin Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Lymphoblastic Lymphoma; Stage I Childhood Small Noncleaved Cell Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Multiple Myeloma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage II Childhood Anaplastic Large Cell Lymphoma; Stage II Childhood Hodgkin Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Childhood Lymphoblastic Lymphoma; Stage II Childhood Small Noncleaved Cell Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Childhood Anaplastic Large Cell Lymphoma; Stage III Childhood Hodgkin Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Lymphoblastic Lymphoma; Stage III Childhood Small Noncleaved Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Multiple Myeloma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage IV Childhood Anaplastic Large Cell Lymphoma; Stage IV Childhood Hodgkin Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Lymphoblastic Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; T-cell Large Granular Lymphocyte Leukemia; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Immunoblastic Lymphadenopathy; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Polycythemia Vera; Primary Myelofibrosis; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (WAITLIST CONTROL GROUP) (Active Comparator): Patients and caregivers receive standard of care and are offered the massage intervention after 8 weeks.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Procedure: standard follow-up care
- Arm II (TOUCH) (Experimental): Caregivers undergo a 60-minute training session on simple massage techniques, including the "Massage Toolkit," comprising Swedish Massage and Trigger Point Therapy Massage, at week 0 and a booster 60-minute massage training session at week 4 with a licensed massage therapist. Caregivers are instructed to massage their children for at least 3 20-minute sessions per week for 8 weeks.
  Interventions: Procedure: massage therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: intervention by caregiver
- Arm III (TOUCH+) (Experimental): Caregivers undergo a 60-minute training session on simple massage techniques, including the "Massage Toolkit," comprising Swedish Massage and Trigger Point Therapy Massage, at week 0 and a booster 60-minute massage training session at week 4 with a licensed massage therapist. Caregivers are instructed to massage their children for at least 3 20-minute sessions per week for 8 weeks. Caregivers also receive a 45-minute massage by the massage therapist.
  Interventions: Procedure: massage therapy; Other: questionnaire administration; Procedure: quality-of-life assessment; Other: intervention by caregiver

INTERVENTIONS:
Procedure: massage therapy — Undergo massage therapy
  Other Names: massage; therapeutic massage
  Arms: Arm II (TOUCH); Arm III (TOUCH+)
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: intervention by caregiver — Undergo massage by caregiver
  Arms: Arm II (TOUCH); Arm III (TOUCH+)
Procedure: standard follow-up care — Undergo standard follow-up care
  Arms: Arm I (WAITLIST CONTROL GROUP)

SUMMARY:
This clinical trial studies massage therapy given by caregiver in treating quality of life of young patients undergoing treatment for cancer. Massage therapy given by a caregiver may improve the quality of life of young patients undergoing treatment for cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and acceptability of conducting a massage intervention with childhood cancer patients and their primary caregivers.

II. To investigate feasibility of implementing a brief targeted massage training protocol with caregivers.

III. To identify barriers to recruitment, intervention adherence, and full study completion by consented families.

IV. To assess preliminary effectiveness of the massage intervention in reducing caregiver and child psychological distress (anxiety, depression, parenting stress) and promoting child health-related quality of life.

V. To compare outcome data between two intervention arms (TOUCH: child massage only; TOUCH+: Caregiver massage plus child massage) and between each arm and a wait list control condition.

VI. To utilize the pilot data in a development of contextually specific and targeted grant application for a fully powered randomized controlled trial of the efficacy of caregiver massage of children undergoing treatment for cancer.

SECONDARY OBJECTIVES:

I. To investigate reciprocal change in self-reported psychosocial functioning within the caregiver-child dyad from baseline to post-intervention.

II. To assess impact of massage intervention upon levels of a stress biomarker (cortisol) in caregivers and children and to assess associations of cortisol levels with self-reported psychosocial functioning.

OUTLINE: Patients and their caregivers are randomized to 1 of 3 treatment arms.

ARM I (WAITLIST CONTROL GROUP): Patients and caregivers receive standard of care and are offered the massage intervention after 8 weeks.

ARM II (TOUCH): Caregivers undergo a 60-minute training session on simple massage techniques, including the "Massage Toolkit," comprising Swedish Massage and Trigger Point Therapy Massage, at week 0 and a booster 60-minute massage training session at week 4 with a licensed massage therapist. Caregivers are instructed to massage their children for at least 3 20-minute sessions per week for 8 weeks.

ARM III (TOUCH+): Caregivers undergo a 60-minute training session on simple massage techniques, including the "Massage Toolkit," comprising Swedish Massage and Trigger Point Therapy Massage, at week 0 and a booster 60-minute massage training session at week 4 with a licensed massage therapist. Caregivers are instructed to massage their children for at least 3 20-minute sessions per week for 8 weeks. Caregivers also receive a 45-minute massage by the massage therapist.

Patients complete questionnaires at weeks 0, 8, and 16.

After completion of study treatment, patients and caregivers are followed for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

Signed protocol specific informed consent by the child's caregiver Assent by the child Caregiver is at least 18 years of age The child is currently treated for cancer (chemotherapy alone, radiation therapy alone, chemotherapy and radiation therapy, chemotherapy and surgery, or radiation therapy and surgery) at Wake Forest Baptist Health (WFBH) Pediatric Oncology The child has at least 16 weeks remaining on their treatment regimen The caregiver and child understand written and spoken English The child has no medical or functional contraindications reported by his/her attending\physician

Exclusion Criteria:

Parents/caregivers who have previously provided consistent massage for their child will be excluded from the study Child is receiving radiation only

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of conducting a massage intervention with childhood cancer patients and their primary caregivers | Up to 16 weeks

SECONDARY OUTCOMES:
Effectiveness of caregiver massage to reduce child and caregiver distress and promote child health-related quality of life | Baseline
Effectiveness of caregiver massage to reduce child and caregiver distress and promote child health-related quality of life | Week 8
Effectiveness of caregiver massage to reduce child and caregiver distress and promote child health-related quality of life | Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Janet Tooze, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States